CLINICAL TRIAL: NCT00606216
Title: Structural Imaging and Cognitive Functions in Adult Stem Cell Transplant Recipients Treated With Chemotherapy Alone or in Combination With Radiotherapy
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 06-162
Record Dates: First submitted 2008-01-21; First posted 2008-02-01 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia; Acute Undifferentiated Leukemia; Biphenotypic Leukemia; Myelodysplastic Syndrome; Non-Hodgkin's Lymphoma
Keywords: MRI
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Biphenotypic, Acute; Myelodysplastic Syndromes; Lymphoma, Non-Hodgkin | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- A: TBI and Chemotherapy Conditioning Regimen. Twenty (20) patients will undergo conditioning treatment with TBI and chemotherapy prior to receiving a myeloablative allogeneic or an autologous HSCT.
  Interventions: Procedure: MRI and cognitive evaluation
- B: Chemotherapy Alone Conditioning Regimen Twenty (20) patients will undergo conditioning treatment with an all chemotherapy regimen prior to receiving an allogeneic or an autologous HSCT.
  Interventions: Procedure: MRI and cognitive evaluation
- C: A cohort of twenty (20) healthy controls, frequency matched on age, gender, and education, will be recruited at WCMC to participate in the study.
  Interventions: Procedure: brain MRI study and a brief neuropsychological evaluation

INTERVENTIONS:
Procedure: MRI and cognitive evaluation — Patients will undergo a brain MRI study and a brief neuropsychological evaluation, at the time of enrollment for controls and prior to undergoing the conditioning treatment required for the stem cell transplant for patients. A follow-up MRI and cognitive evaluation will be performed approximately 12 months after the transplant for patients.
  Groups: A
Procedure: MRI and cognitive evaluation — Pt will undergo a Magnetic Resonance Imaging (MRI) study of the brain and a brief neuropsychological evaluation, at the time of enrollment for healthy controls and prior to undergoing the conditioning treatment required for the stem cell transplant for patients (Baseline/Time 1).
  Groups: B
Procedure: brain MRI study and a brief neuropsychological evaluation — A brain MRI study and a brief neuropsychological evaluation will be performed at baseline (Time 1). A follow-up MRI and cognitive evaluation will be performed and about 12 months after the baseline for healthy controls
  Groups: C

SUMMARY:
The purpose of this study is to learn about possible changes in brain anatomy and in thinking abilities, such as memory skills, in patients with cancer who receive treatment with chemotherapy alone or in combination with total body radiation before undergoing stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with acute myeloid leukemia (AML), acute lymphoblastic leukemia (ALL), acute undifferentiated or biphenotypic leukemia, myelodysplastic syndrome (MDS), Hodgkin's lymphoma, (HL) or non-Hodgkin's lymphoma (NHL), and in complete remission at the time of enrollment
* Are scheduled to undergo conditioning treatment with (1) total body radiation (TBI) and chemotherapy or (2) chemotherapy alone prior to receiving a myeloablative allogeneic HSCT
* Between 18 and 70 years of age.
* Are English speaking.
* Have capacity to give consent.

Healthy Control Inclusion Criteria:

* Have no diagnosis of cancer except basal cell carcinoma
* Between 18 and 70 years of age.
* Are English speaking.
* Have capacity to give consent

Exclusion Criteria:

* Patients with signs and/or symptoms of central nervous system disease as determined by their physician or by a brain MRI, either at the time of enrollment or during the study period.
* With disease progression at the time of enrollment or during the study period
* With self-reported Axis I psychiatric disorder (DSM-IV), major affective disorder (untreated), bipolar disorder, schizophrenia
* With a history of a neurological disorder, neurodegenerative disease, or traumatic brain injury with loss of consciousness
* With standard contraindications to MRI examinations

Healthy Control Exclusion Criteria:

* Exposure to chemotherapy or radiation therapy for any medical condition
* With self-reported Axis I psychiatric disorder (DSM-IV), major affective disorder (untreated), bipolar disorder, schizophrenia
* With a history of neurological disorders, neurodegenerative disease, or traumatic brain injury with loss of consciousness
* With standard contraindications to MRI examinations

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be identified and recruited to participate in the study by Memorial Sloan-Kettering Cancer Center (MSKCC) and Weill Cornell Medical Center (WCMC).
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2007-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
assess changes in hippocampal volume & white matter integrity prospectively in adult ca pts who get treatment w/i chemotherapy alone or in combination with total body irradiation (TBI) before undergoing hematopoietic stem cell transplantation. | conclusion of the study

SECONDARY OUTCOMES:
assess memory and executive functions prospectively in these patients. We will investigate whether there is an association between structural brain changes and cognitive performance. | conclusion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Denise Correa, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medical Center, New York, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org